CLINICAL TRIAL: NCT03234374
Title: A Randomized, Single Blind Study to Investigate the PK, Relative Bioavailability and Safety of INL-001 Bupivacaine HCl Collagen-Matrix Implant 300 mg Compared to Marcaine™ 0.25% (Bupivacaine HCl) 175 mg Infiltration After Open Hernioplasty
Brief Title: Pharmacokinetics, Relative Bioavailability and Safety of INL-001 Compared to Marcaine After Open Hernioplasty
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Innocoll (Industry)
Collaborators: Medpace, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: INN-CB-022
Record Dates: First submitted 2017-06-28; First posted 2017-07-31 (Actual); Results first posted 2020-12-31 (Actual); Last update posted 2021-07-30 (Actual); Status verified 2021-07

CONDITIONS: Hernioplasty
Keywords: Pharmacokinetics; Bioavailability; Safety; Bupivacaine; Collagen; Implant; Marcaine; Hernioplasty
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant
Masking Description: This is a single-blind study in which the study subject is blinded to treatment group. All precautions will be taken to ensure that the blinding of the treatment group is maintained throughout the study period. Unblinding to the subject will not be permitted unless it is deemed necessary for appropriate treatment of a medical emergency.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- INL-001 (Experimental): 3 x 100 mg INL-001 (bupivacaine HCl collagen implants). Total bupivacaine HCl dose 300 mg.
  Interventions: Combination Product: INL-001 (bupivacaine HCl collagen implant)
- Marcaine 0.25% infiltration (Active Comparator): Marcaine 0.25% infiltration (bupivacaine HCl 175 mg).
  Interventions: Drug: Marcaine 0.25% infiltration

INTERVENTIONS:
Combination Product: INL-001 (bupivacaine HCl collagen implant) — 3 x 100 mg INL-001 bupivacaine HCl collagen-matrix implants (total bupivacaine HCl dose 300 mg)
  Other Names: INL-001
  Arms: INL-001
Drug: Marcaine 0.25% infiltration — Marcaine 0.25% (bupivacaine HCl) 175 mg infiltration
  Other Names: Marcaine
  Arms: Marcaine 0.25% infiltration

SUMMARY:
This is a multicenter randomized, single-blind, controlled study. The primary objectives of this study are to obtain the pharmacokinetic profile and the relative bioavailability of the INL-001 matrix during and after open hernioplasty compared to Marcaine™ 0.25% infiltration.

DETAILED DESCRIPTION:
This is a multicenter randomized, single-blind, controlled study. Prior to surgery on Day 1, 48 subjects who continue to meet study entry criteria will be randomized just prior to surgery in a 2:1 ratio to receive either 3 x 100 mg INL-001 bupivacaine HCl collagen-matrix implants (total bupivacaine HCl dose 300 mg) or Marcaine 0.25% (bupivacaine HCl) 175 mg infiltration. Subjects will then undergo open hernioplasty according to standard procedure.

Subjects will remain in the clinic at least until after the 72 hour blood sample has been collected for PK analysis on Day 4. Subjects discharged after the 72 hour blood draw will be instructed to return to the clinic to complete the 96 hour PK blood draw on Day 5. Follow-up safety assessments will include clinic visits on Day 7, Day 15 and Day 30.

Pharmacokinetic blood samples will be collected from subjects before surgery and at predetermined time points up to 96 hours after administration of study drug. Safety assessments will include frequent assessment of vital signs through 72 hours, continuous electrocardiogram (ECG) monitoring for at least 24 hours, oxygen saturation levels, and adverse events (AEs) reporting with particular emphasis on the signs and symptoms of CNS and cardiovascular bupivacaine toxicity. The surgical wound will be assessed frequently for adverse events associated with altered wound healing.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for inclusion into the study, subjects must:

* Be a man or woman ≥18 years of age.
* Be eligible for unilateral inguinal hernioplasty with mesh (open laparotomy, tension-free technique) performed according to standard surgical technique under general anesthesia. Repair of multiple hernias through a single incision is permitted. If female of childbearing potential, have a negative pregnancy test at screening and before randomization on Day 1 AND be using an effective contraception method (ie, abstinence, intrauterine device [IUD], hormonal [estrogen/progestin] contraceptives, or barrier control) for at least one menstrual cycle prior to study enrollment and for the duration of the study, OR be surgically sterile, OR be a postmenopausal female (no menses for at least 1 year or hysterectomy).
* Has the ability and willingness to comply with the study procedures.
* Be willing to use only permitted medications throughout the study.
* Be willing to use opioid analgesia.
* Be able to fluently speak and understand either English or Spanish and be able to provide meaningful written informed consent for the study.

Exclusion Criteria:

A subject will be excluded from study participation if prior to surgery he/she:

* Has a known hypersensitivity to amide local anesthetics, morphine, acetaminophen, or bovine products.
* Is scheduled for bilateral inguinal hernioplasty or other significant concomitant surgical procedure.
* Has undergone major surgery within 3 months of the scheduled hernioplasty or plans to undergo another laparotomy procedure within the 30 day postoperative period.
* Has known or suspected history of alcohol or drug abuse or misuse within 3 years of screening or evidence of tolerance or physical dependency on opioid analgesics or sedative-hypnotic medications.
* Has any clinically significant unstable cardiac, neurological, immunological, renal, hepatic or hematological disease or any other condition that, in the opinion of the investigator, could compromise the subject's welfare, ability to communicate with the study staff or otherwise contraindicate study participation.
* Has venous access difficulties that may preclude the frequent pharmacokinetic sampling requirements of the study.
* Has participated in a clinical trial (investigational or marketed product) within 30 days of surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2017-06-02 (Actual); Primary Completion 2017-08-15 (Actual); Study Completion 2017-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gwendolyn Niebler, D.O., Study Director — Innocoll
Locations (5):
- United States (5):
  - Pinnacle Research Group, Anniston, Alabama
  - Park Place Surgery Center, Longwood, Florida
  - Research Concepts, Houston, Texas
  - Research Concepts GP, LLC - Houston, Houston, Texas
  - Jean Brown Research, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Leiman D, Niebler G, Minkowitz HS. Pharmacokinetics and Safety of INL-001 (Bupivacaine HCl) Implants Compared with Bupivacaine HCl Infiltration After Open Unilateral Inguinal Hernioplasty. Adv Ther. 2021 Jan;38(1):691-706. doi: 10.1007/s12325-020-01565-x. Epub 2020 Nov 25. PMID 33237534

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | INL-001 | Marcaine 0.25% Infiltration
Started | 35 | 17
Completed | 34 | 16
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Population: Safety & PK Population
Groups:
- Total: Total of all reporting groups
Arm/Group | INL-001 | Marcaine 0.25% Infiltration | Total
Number analyzed (Participants) | 34 | 16 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.6 (14.84) | 41.6 (12.18) | 44.3 (14.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 33 | 16 | 49
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 3 | 0 | 3
  White | 31 | 15 | 46
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 34 | 16 | 50

OUTCOME MEASURES:

1. Primary Outcome: Cmax
Description: Maximum (peak) plasma concentration
Time Frame: 0.5, 1, 1.5, 2, 3, 4, 5, 6, 9, 12, 18, 24, 36, 48 and 72 hours.
Population: Per-Protocol PK Population
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | INL-001 | Marcaine 0.25% Infiltration
Number analyzed (Participants) | 34 | 16
ng/ml | 663.412 (263.826) | 641.000 (262.684)

2. Primary Outcome: Tmax
Description: Time to maximum (peak) plasma concentration
Time Frame: 0.5, 1, 1.5, 2, 3, 4, 5, 6, 9, 12, 18, 24, 36, 48 and 72 hours
Population: Summary of Plasma Bupivacaine PK Parameters by Treatment - Per-Protocol PK Population
Measure: Median (Full Range); unit: hours
Arm/Group | INL-001 | Marcaine 0.25% Infiltration
Number analyzed (Participants) | 34 | 16
hours | 3.03 [1.48 to 24.02] | 1.01 [0.53 to 3.97]

3. Primary Outcome: Tlag
Description: Lag-time
Time Frame: 0.5, 1, 1.5, 2, 3, 4, 5, 6, 9, 12, 18, 24, 36, 48 and 72 hours
Population: Per-Protocol PK Population
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | INL-001 | Marcaine 0.25% Infiltration
Number analyzed (Participants) | 34 | 16
hours | 0.51 (0.13) | 0.47 (0.13)

4. Primary Outcome: t½ Terminal Half Life
Description: Terminal half-life
Time Frame: 0.5, 1, 1.5, 2, 3, 4, 5, 6, 9, 12, 18, 24, 36, 48 and 72 hours
Population: Per-Protocol PK Population
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | INL-001 | Marcaine 0.25% Infiltration
Number analyzed (Participants) | 34 | 16
hours | 0.04 (0.01) | 0.09 (0.04)

5. Primary Outcome: λz
Description: Terminal phase rate constant
Time Frame: 0.5, 1, 1.5, 2, 3, 4, 5, 6, 9, 12, 18, 24, 36, 48 and 72 hours
Population: Per protocol population
Measure: Mean (Standard Deviation); unit: 1/hour
Arm/Group | INL-001 | Marcaine 0.25% Infiltration
Number analyzed (Participants) | 34 | 16
1/hour | 18.95 (5.95) | 9.08 (3.75)

6. Primary Outcome: AUC
Description: Area under the plasma concentration-time curve from Time 0 to last time of last quantifiable plasma concentration (AUC0-last)
Time Frame: 0.5, 1, 1.5, 2, 3, 4, 5, 6, 9, 12, 18, 24, 36, 48 and 72 hours
Population: Per Protocol Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/[mL*mg]
Arm/Group | INL-001 | Marcaine 0.25% Infiltration
Number analyzed (Participants) | 34 | 16
h*ng/[mL*mg] | 18,186.9 (39.0) | 8836.9 (46.3)

7. Primary Outcome: AUC0-∞
Description: AUC from Time 0 to infinity
Time Frame: 0.5, 1, 1.5, 2, 3, 4, 5, 6, 9, 12, 18, 24, 36, 48 and 72 hours
Population: Per protocol population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/[mL*mg]
Arm/Group | INL-001 | Marcaine 0.25% Infiltration
Number analyzed (Participants) | 34 | 16
h*ng/[mL*mg] | 19,012.5 (38.7) | 8920.1 (0.65)

8. Primary Outcome: AUC Extrapolated
Description: AUC = area under the plasma concentration-time curve;
Time Frame: 0.5, 1, 1.5, 2, 3, 4, 5, 6, 9, 12, 18, 24, 36, 48 and 72 hours
Measure: Geometric Mean (Standard Deviation); unit: (h*ng/mL)
Arm/Group | INL-001 | Marcaine 0.25% Infiltration
Number analyzed (Participants) | 34 | 16
(h*ng/mL) | 2.96 (120.9) | 0.65 (122.5)

ADVERSE EVENTS:
Time Frame: 30 days
Description: Safety Population
Arm/Group | INL-001 | Marcaine 0.25% Infiltration
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/16
Other Adverse Events (participants affected / at risk) | 33/34 | 15/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | INL-001 (N=34) | Marcaine 0.25% Infiltration (N=16)
Somnolence (Nervous system disorders) | 19 (19) | 10 (10)
Dizziness (Nervous system disorders) | 12 (12) | 7 (7)
Tremor (Nervous system disorders) | 6 (6) | 3 (3)
Dysgeusia (Nervous system disorders) | 4 (4) | 4 (4)
Headache (Nervous system disorders) | 4 (4) | 1 (1)
Constipation (Gastrointestinal disorders) | 8 (8) | 1 (1)
Hypoaesthesia oral (Gastrointestinal disorders) | 3 (3) | 2 (2)
Nausea (Gastrointestinal disorders) | 3 (3) | 2 (2)
Paraesthesia oral (Gastrointestinal disorders) | 3 (3) | 2 (2)
Vision blurred (Eye disorders) | 8 (8) | 3 (3)
Restlessness (Psychiatric disorders) | 6 (6) | 2 (2)
Anxiety (Psychiatric disorders) | 2 (2) | 1 (1)
Incision site complication (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 3 (3) | 1 (1)
Bradycardia (Cardiac disorders) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-17): https://cdn.clinicaltrials.gov/large-docs/74/NCT03234374/Prot_SAP_000.pdf